CLINICAL TRIAL: NCT00950274
Title: Intramyocardial Transplantation of Bone Marrow Stem Cells for Improvement of Post-infarct Myocardial Regeneration in Addition to CABG Surgery: a Controlled, Prospective, Randomized, Double Blinded Multicenter Trial (PERFECT)
Brief Title: Intramyocardial Transplantation of Bone Marrow Stem Cells in Addition to Coronary Artery Bypass Graft (CABG) Surgery
Acronym: PERFECT
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Recruitment stopped due to slow recruitment
Sponsor: Miltenyi Biotec B.V. & Co. KG (Industry)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Responsible Party: Sponsor
Organization: Miltenyi Biomedicine GmbH (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PERFECT 001; M-2006-144 (Other: Sponsor)
Record Dates: First submitted 2009-07-30; First posted 2009-07-31 (Estimated); Last update posted 2020-07-15 (Actual); Status verified 2018-08

CONDITIONS: Myocardial Ischemia; Coronary Artery Disease
Keywords: Cell therapy; Bone marrow; CD133; Bypass surgery; Stem cells; Myocardial infarction; Myocardial ischemia
MeSH Terms: conditions — Myocardial Ischemia; Coronary Artery Disease; Myocardial Infarction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CD133+ autologous bone marrow stem cells (Active Comparator)
  Interventions: Drug: CD133+ autologous bone marrow stem cell
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CD133+ autologous bone marrow stem cell — Intramyocardial injection of 5 mL CD133+ cells (0.5-5x10e6 cells) suspended in physiological saline + 10% autologous serum intramyocardially during CABG surgery
  Arms: CD133+ autologous bone marrow stem cells
Drug: Placebo — Intramyocardial injection of 5 mL of physiological saline + 10% autologous serum intramyocardially during CABG surgery
  Arms: Placebo

SUMMARY:
In spite of the fact that the post-myocardial infarction survival rate has improved with recent medical advances, reduced heart function attributed to irreversible loss of viable cardiomyocytes is still a major clinical problem.

The aim of the current study is to determine whether intramyocardial injection of autologous CD133+ bone marrow stem cells yields a functional benefit in addition to coronary artery bypass graft (CABG) surgery in patients with chronic ischemic coronary artery disease.

DETAILED DESCRIPTION:
Beginning in 2001, a phase-1 equivalent feasibility and safety evaluation of intramyocardial injection of autologous CD133+ bone marrow cells during elective CABG surgery was conducted at Rostock University. No procedure-related adverse events were observed and there was some improvement of myocardial contractility and perfusion. It was decided to proceed with a controlled efficacy testing, comparing the outcome of standard CABG surgery with that after CABG and CD133+ cell injection. The results of that study indicate that the additional cell injection yields a better left ventricular contractility than CABG alone (LVEF = 47.1±8% vs. 41.3±9% at 6 months). Although this result is encouraging, the trial had several limitations that hamper interpretation of the data. Most notably, no sham-injection of placebo material was performed in the control group, and standard 2D echocardiography served as the only measurement of global LV contractility.

However, there were no procedure-related complications up to 18 months postoperatively, especially no new ventricular arrhythmia or neoplasia.

Therefore, a prospective, double blinded, randomized, and placebo-controlled multi-center trial will be conducted in Germany, employing current state-of-the art measurement of global and regional LV contractility by cardiac MRI. The following hypothesis will be tested: "Patients who undergo CABG & CD133+ cell injection do not have a higher LV ejection fraction than patient who undergo CABG alone, measured 6 months after the operation". A power analysis based on the previous trial results indicated that 71 patients per group need to be enrolled so as to reject the null-hypothesis with sufficient statistical power. A total of 142 patients will therefore be enrolled in the study. Patients will be randomized in a 1:1 ratio to undergo CABG surgery in conjunction with either intramyocardial injection of autologous CD133-enriched bone marrow cells or placebo. Bone marrow will be harvested one or two days prior to surgery and a CD133-enriched cell product (or placebo) will be prepared at a central cell processing GMP unit. Bypass surgery will be performed and the investigational product will be injected in the border zone of the infarcted myocardium. Random allocation will be performed in the cell production facility, so that neither the patient nor the surgeon nor any of the personnel involved in follow-up examinations will know whether the cell product or placebo was administered. The primary outcome parameter (LVEF at 6 months) will be measured by cardiac MRI, and secondary outcome parameters include physical exercise capacity, cardiac function, safety and Quality of Life (QoL).

ELIGIBILITY:
Inclusion Criteria:

* Coronary artery disease after myocardial infarction with indication for CABG surgery
* Currently reduced global LVEF assessed at site by cardiac MRI at rest (25% ≤ LVEF ≤ 50%)
* Presence of a localized akinetic/hypokinetic/hypoperfused area of LV myocardium for defining the target area
* Informed consent of the patient
* 18 years ≤ Age < 80 years
* Are not pregnant and do not plan to become pregnant during the study. Females with childbearing potential must provide a negative pregnancy test within 1-7 days before OP and must be using oral or injectable contraception (non-childbearing potential is defined as post-menopausal for at least 1 year or surgical sterilization or hysterectomy at least 3 months before study start).

Exclusion Criteria:

* Emergency operation
* Presence of any moderate-severe valvular heart disease requiring concomitant valve replacement or reconstruction
* Medical History of recent resuscitation in combination with ventricular arrhythmia classified by LOWN ≥ class II
* Acute myocardial infarction within last 2 weeks
* Debilitating other disease: Degenerative neurologic disorders, psychiatric disease, terminal renal failure requiring dialysis, previous organ transplantation, active malignant neoplasia, or any other serious medical condition that, in the opinion of the Investigator is likely to alter the patient's course of recovery or the evaluation of the study medication's safety
* Impaired ability to comprehend the study information
* Absent informed written consent
* Treatment with any investigational drug within the previous 30 days
* Apparent infection (c-reactive protein [CRP] ≥ 20 mg/L, fever ≥ 38.5° C)
* Contraindication for MRI scan
* Immune compromise including active infection with Hepatitis B, C, HIV virus or seropositivity for Treponema pallidum
* Pregnant or breast feeding
* Childbearing potential with unreliable birth control methods
* Have previously been enrolled in this study, respectively phase I and phase II
* Known hypersensitivity or sensitization against murine products and human-anti-mouse-antibody-titer ≥ 1:1000
* Contraindication to bone marrow aspiration
* Known hypersensitivity against iron dextran

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2009-07; Primary Completion 2016-03 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Left ventricular ejection fraction at rest, measured by MRI | 6 months

SECONDARY OUTCOMES:
Change in LVEF as assessed by MRI and echocardiography | early postoperatively and 6 months
Regional contractility in the AOI / Change in LV dimensions (left ventricular end systolic diameter [LVESD], left ventricular end diastolic diameter [LVEDD]) as assessed by echocardiography | early postoperatively (discharge), 6 months
Physical exercise capacity determined by 6 minute walk test | early postoperatively (discharge), 6 months
NYHA and CCS class | early postoperatively (discharge), 6 months
MACE (cardiac death, myocardial infarction, secondary intervention/reoperation, ventricular arrhythmia) | 6 months
QoL-score: Minnesota Living with Heart Failure Questionnaire, SF36 Questionnaire, EQ-5D Questionnaire | 3 months, 6 months post-OP

CONTACTS AND LOCATIONS:
Overall Officials: Gustav Steinhoff, M.D., Principal Investigator — Universitiy of Rostock
Locations (6):
- Germany (6):
  - Herz- und Diabeteszentrum Nordrhein Westfalen, Bad Oeynhausen
  - Deutsches Herzzentrum Berlin, Berlin
  - Universitäres Herzzentrum Hamburg, Hamburg
  - Medical School Hannover, Hanover
  - Herzzentrum Universität Leipzig, Leipzig
  - University of Rostock, Rostock

REFERENCES:
- [Derived] Wolfien M, Klatt D, Salybekov AA, Ii M, Komatsu-Horii M, Gaebel R, Philippou-Massier J, Schrinner E, Akimaru H, Akimaru E, David R, Garbade J, Gummert J, Haverich A, Hennig H, Iwasaki H, Kaminski A, Kawamoto A, Klopsch C, Kowallick JT, Krebs S, Nesteruk J, Reichenspurner H, Ritter C, Stamm C, Tani-Yokoyama A, Blum H, Wolkenhauer O, Schambach A, Asahara T, Steinhoff G. Hematopoietic stem-cell senescence and myocardial repair - Coronary artery disease genotype/phenotype analysis of post-MI myocardial regeneration response induced by CABG/CD133+ bone marrow hematopoietic stem cell treatment in RCT PERFECT Phase 3. EBioMedicine. 2020 Jul;57:102862. doi: 10.1016/j.ebiom.2020.102862. Epub 2020 Jul 4. PMID 32629392
- [Derived] Steinhoff G, Nesteruk J, Wolfien M, Kundt G; PERFECT Trial Investigators Group; Borgermann J, David R, Garbade J, Grosse J, Haverich A, Hennig H, Kaminski A, Lotz J, Mohr FW, Muller P, Oostendorp R, Ruch U, Sarikouch S, Skorska A, Stamm C, Tiedemann G, Wagner FM, Wolkenhauer O. Cardiac Function Improvement and Bone Marrow Response -: Outcome Analysis of the Randomized PERFECT Phase III Clinical Trial of Intramyocardial CD133+ Application After Myocardial Infarction. EBioMedicine. 2017 Aug;22:208-224. doi: 10.1016/j.ebiom.2017.07.022. Epub 2017 Jul 29. PMID 28781130
- [Derived] Donndorf P, Kaminski A, Tiedemann G, Kundt G, Steinhoff G. Validating intramyocardial bone marrow stem cell therapy in combination with coronary artery bypass grafting, the PERFECT Phase III randomized multicenter trial: study protocol for a randomized controlled trial. Trials. 2012 Jul 2;13:99. doi: 10.1186/1745-6215-13-99. PMID 22747980